CLINICAL TRIAL: NCT00655460
Title: Clinical Process Improvement With A Bedside Computerized Insulin Therapy Protocol For Blood Glucose Control (eProtocol-insulin) in Adult And Pediatric ICU Patients:Further Refinement and Validation of eProtocol-insulin
Brief Title: Improving Blood Glucose Control With a Computerized Decision Support Tool: Phase 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01-HC-45210-1; HHSN268200425210C
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2008-01

CONDITIONS: Critically Ill; Hyperglycemia
Keywords: Glucose; Insulin; computer; critical care
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eProtocol (Experimental)
  Interventions: Procedure: glucose control with computer generated recommendations

INTERVENTIONS:
Procedure: glucose control with computer generated recommendations — Insulin dosing will be recommended by the computer tools based on subject glucose values. Bedside clinicians will have the ablity to accept or reject the suggested dose.

SUMMARY:
The Purpose of this study is to:

1. Refine and validate a computerized bedside decision support tool blood glucose management in critically ill adult and pediatric ICU patients.
2. Monitor how often low blood sugar levels occur during use of the bedside tool.
3. Determine how the computerized tool effects the workload of the ICU nurses.

DETAILED DESCRIPTION:
This first phase will be a prospective cohort study. We will validate the bedside tool in at least 4 adult and at least 4 pediatric ICUs and if necessary we will modify the bedside tool. The computerized bedside tool will be considered refined if >90% of the generated instructions are accepted and if the percent of glucose values in the 70-110 mg/dl range are equivalent to our pilot experience rate of 55%, and if the rate of glucose values less than or equal to 40 mg/dl is less than 0.5% of glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric ICU: Proposed indications by pediatric clinicians at participating ICUs for glucose control in their ICUs would include patients who require mechanical ventilation for greater than 24 hours and/or require a vasoactive infusion (e.g. dopamine >3 mg/kg/min, dobutamine, epinephrine, or vasopressin).
2. Adult ICUs: Proposed indications by clinicians in participating ICUs for glucose control in participating adult ICUs include critically ill patients with an anticipated ICU length of stay of 3 or more days.

Exclusion Criteria:

1. Pregnancy (negative pregnancy test required for females of child-bearing age)
2. Age less than one month
3. Inborn errors of metabolism that the clinician suspects will affect glucose homeostasis
4. Acute or chronic liver disease with any documented episode of blood or plasma glucose <60 mg/dl within the 24 hours prior to study entry
5. Diabetic Ketoacidosis (critically ill patients with insulin dependent diabetes not in ketoacidosis will be eligible if attending physicians intend to use intravenous insulin as part of ordinary care)
6. Severe chronic liver disease (Child-Pugh score >10)

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable during Phase I will be the acceptability of the eProtocol-insulin instructions (compliance of bedside clinicians with instructions: more than 90 % of all instructions accepted by the bedside clinician). | 3 years

SECONDARY OUTCOMES:
Proportion of glucose determinations within the range of 70-110 mg/dl (3.9-6.1 mMol/l) | 3 years
Nursing perception of workload in comparison to ordinary care | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Morris, MD, Principal Investigator — Intermountain Medical Center, Murray, Utah
Locations (11):
- United States (11):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Pennsylvania State Children's Hospital, Hersey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - LDS Hospital, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia